CLINICAL TRIAL: NCT06437145
Title: Acute Effects of High Intensity Interval Training (HIIT) vs. Moderate Intensity Continuous Training (MICT) on Heart Rate Variability Parameters in Patients After Myocardial Infarction
Brief Title: Acute Effects of HIIT vs. MICT on HRV
Acronym: MW2acute
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Borut Jug, Prof., University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UKCLRehab2024/1
Record Dates: First submitted 2024-04-16; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction
Keywords: exercise training; high intensity interval training; moderate intensity continuous training; heart rate variability; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Each patient will have a bout of HIIT during one session and a bout of MICT during another session performed in a random order.
Who Masked: Outcomes Assessor
Masking Description: HRV parameters analysis will be blinded regarding the exercise training modality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (HIIT) (Active Comparator): The high-intensity interval training session consists of 5-min warm-up and 5-min cool-down periods. The main part has 7 cycles. Each cycle consists of 1.5 min of 80-90% of HRpeak and 3 min of 65-70% of HRpeak.
  Interventions: Other: Type of Exercise
- Moderate intensity continuous training (MICT) (Active Comparator): The moderate-intensity continuous training session consists of 5 min warm-up and 3-min cool down period. The main part consists of 32 min of 75% of HRpeak.
  Interventions: Other: Type of Exercise

INTERVENTIONS:
Other: Type of Exercise — The high-intensity interval training session consists of 5-min warm-up and 5-min cool-down periods. The main part has 7 cycles. Each cycle consists of 1.5 min of 80-90% of HRpeak and 3 min of 65-70% of HRpeak. The moderate-intensity continuous training session consists of 5 min warm-up and 3-min cool down period. The main part consists of 32 min of 75% of HRpeak.

SUMMARY:
Heart rate variability (HRV) is impaired in patients after myocardial infarction. Most studies so far have proved chronic beneficial effects of different types of exercise on HRV parameters. Data on acute effects of different types of exercise training (e.g. high intensity interval training [HIIT] and moderate intensity continuous training [MICT]) is scarce.

Patients in the study will perform both HIIT and MICT in a random order and in-between break of at least 48 hours. A 5-minute high resolution ECG recording will be performed before and immediately after both HIIT and MICT.

ELIGIBILITY:
Inclusion Criteria:

* myocardial infarction in last 120 days
* sinus rhythm

Exclusion Criteria:

* contraindications for exercise training
* uncontrolled dysrhythmias
* Heart Failure NYHA IV stage
* cognitive impairment
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
HF parameter | 5-minutes high resolution ECG recording before and after an exercise session
  High frequency domain of the HRV

SECONDARY OUTCOMES:
LF parameter | 5-minutes high resolution ECG recording before and after an exercise session
  Low frequency domain of the HRV
SDNN | 5-minutes high resolution ECG recording before and after an exercise session
  Standard deviation of NN intervals
RMSSD | 5-minutes high resolution ECG recording before and after an exercise session
  Root mean square of successive RR interval differences
pNN50 | 5-minutes high resolution ECG recording before and after an exercise session
  Percentage of successive RR intervals that differ by more than 50 ms

OTHER OUTCOMES:
Non-linear methods | 5-minutes high resolution ECG recording before and after an exercise session
  SD1, SD2

CONTACTS AND LOCATIONS:
Overall Officials: Marko Novaković, MD, PhD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Routledge FS, Campbell TS, McFetridge-Durdle JA, Bacon SL. Improvements in heart rate variability with exercise therapy. Can J Cardiol. 2010 Jun-Jul;26(6):303-12. doi: 10.1016/s0828-282x(10)70395-0. PMID 20548976
- [Background] El-Malahi O, Mohajeri D, Mincu R, Bauerle A, Rothenaicher K, Knuschke R, Rammos C, Rassaf T, Lortz J. Beneficial impacts of physical activity on heart rate variability: A systematic review and meta-analysis. PLoS One. 2024 Apr 5;19(4):e0299793. doi: 10.1371/journal.pone.0299793. eCollection 2024. PMID 38578755
- [Background] Grassler B, Thielmann B, Bockelmann I, Hokelmann A. Effects of different exercise interventions on heart rate variability and cardiovascular health factors in older adults: a systematic review. Eur Rev Aging Phys Act. 2021 Nov 17;18(1):24. doi: 10.1186/s11556-021-00278-6. PMID 34789148